CLINICAL TRIAL: NCT03843229
Title: Clinical Trial of Cinobufacini Combined With Transarterial Chemoembolization (TACE) on Primary Liver Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PJ-KS-KY-2018-07(x)
Record Dates: First submitted 2019-02-10; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Liver Cancer
Keywords: Cinobufacini
MeSH Terms: conditions — Liver Neoplasms | interventions — huachansu

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): The treatment group receives Cinobufacini injection 20ml via hepatic artery during Transarterial Chemoembolization(TACE) operation , Cinobufacini injection 20ml+5% Glucose injection 500ml from the second day of TACE until 7th day, and Cinobufacini tablet 3 tablets Tid for 2 months.
  Interventions: Drug: Cinobufacini injection; Procedure: Transarterial Chemoembolization(TACE); Drug: cinobufacini tablet
- control group (Other): The control group only receives Transarterial Chemoembolization (TACE).
  Interventions: Procedure: Transarterial Chemoembolization(TACE)

INTERVENTIONS:
Drug: Cinobufacini injection — The treatment group receives Cinobufacini injection 20ml via hepatic artery during TACE operation , Cinobufacini injection 20ml+5% Glucose injection 500ml from the second day of TACE until 7th day, and Cinobufacini tablet 3 tablets Tid for 2 months.
  Arms: treatment group
Procedure: Transarterial Chemoembolization(TACE) — TACE consists of an injection containing a mixture of chemotherapeutic agents and lipiodol followed by embolization with polyvinyl alcohol (PVA) particles until complete stasis was achieved in the tumor-feeding vessels.Tumor-feeding vessels should be selected/superselected whenever possible.
Drug: cinobufacini tablet — The treatment group receives Cinobufacini injection 20ml via hepatic artery during TACE operation , Cinobufacini injection 20ml+5% Glucose injection 500ml from the second day of TACE until 7th day, and Cinobufacini tablet 3 tablets Tid for 2 months.
  Arms: treatment group

SUMMARY:
The clinical trail of Cinobufacini combined with TACE on primary liver cancer.The trail is randomized controled.Patients are diagnosed primary liver cancer based on pathology or cell biology.They are randomized into 2 groups:both groups receive TACE.The treatment group receives Cinobufacini injection 20ml via hepatic artery during Transarterial Chemoembolization(TACE) operation , Cinobufacini injection 20ml+5% Glucose injection 500ml from the second day of TACE until 7th day, and Cinobufacini tablet 3 tablets Tid for 2 months..The control group only receives TACE.Mainly to study Cinobufacini leads to the influence of the immunologic function after TACE.Immunological examination and Blood biochemistry evaluation include the number ratio、activity and function of immune cell,the immune cell marker(CD3、CD4、CD8,etc),tumor marker(CEA、AFP),etc.Clinical evaluation includes image data(CT/MRI),drug toxicities,quality of life(QOL),etc.

DETAILED DESCRIPTION:
The clinical trail of Cinobufacini combined with TACE on primary liver cancer.The trail is randomized controled.Patients are diagnosed primary liver cancer based on pathology or cell biology.They are randomized into 2 groups:both groups receive TACE.The treatment group receives Cinobufacini injection 20ml via hepatic artery during Transarterial Chemoembolization(TACE) operation , Cinobufacini injection 20ml+5% Glucose injection 500ml from the second day of TACE until 7th day, and Cinobufacini tablet 3 tablets Tid for 2 months..The control group only receives TACE.Mainly to study Cinobufacini leads to the influence of the immunologic function after TACE.Immunological examination and Blood biochemistry evaluation include the number ratio、activity and function of immune cell,the immune cell marker(CD3、CD4、CD8,etc),tumor marker(CEA、AFP),etc.Clinical evaluation includes image data(CT/MRI),drug toxicities,quality of life(QOL),etc.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-70 years.
* male and female.
* signed the informed consent form.
* Diagnosis:Primary liver cancer diagnosed by imaging、cell and pathology report.
* Eastern Cooperative Oncology Group (ECOG) :0-2;life expectancy more than 3 months.
* Indication for TACE,no contraindication.
* First time chemotherapy or at least 6 months after last chemotherapy and radiotherapy.
* At least 8 weeks after last biotherapy.
* Surgery：had not received transplantation surgery,at least 2 weeks after last major surgery.

Exclusion Criteria:

* Chemotherapy is contraindicated.
* Have the primary disease can cause the neuropathy.
* A history of other malignant tumor in recent 5 years.
* Less than 6 months after last chemotherapy or radiotherapy.
* Less than 8 months after last.
* Cinobufacini allergy.
* Had received transplantation surgery ,less than 2 weeks after last major surgery.
* Other researchers think is not suitable for this clinical trail.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-01-27 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
tumor size | the 8th week after TACE operation

SECONDARY OUTCOMES:
the number of CD4+T cell,CD8+T cell in blood | the 8th week after TACE operation
Interleukin(IL)-2,Interleukin(IL)-4,Interleukin(IL)-6,tumor necrosis factor(TNF)-α，interferon(INF)-γ in blood | the 8th week after TACE operation

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD,PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (1):
- The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided